CLINICAL TRIAL: NCT00426010
Title: Measuring Placebo Effect by Elimination and Investigating Its Mechanism of Action
Brief Title: Measuring Placebo Effect by Elimination and Investigating Mechanism of Action
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Collaborators: King AbdulAziz City for Science and Technology (Other)
Responsible Party: Muhammad Hammami, King faisal specialist hospital & research center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RAC# 2051072; KACST:ARP-26-45
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Placebo Effect; Placebo Mechanisms of Action
Keywords: Placebo effect; Caffeine; Systolic BP; VAS
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (4):
- 1 (Active Comparator): overt then covert caffeine
  Interventions: Drug: caffeine/placebo
- 2 (Active Comparator): covert then overt caffeine
  Interventions: Drug: caffeine/placebo
- 3 (Active Comparator): overt then covert placebo
  Interventions: Drug: caffeine/placebo
- 4 (Active Comparator): covert then overt placebo
  Interventions: Drug: caffeine/placebo

INTERVENTIONS:
Drug: caffeine/placebo — caffeine or placebo, either overt or covert

SUMMARY:
We propose to measure the effect of placebo by elimination as well as by a "balanced placebo" design, determine its interaction with active drug, and explore whether placebo exerts part of its effect at the pharmacokinetics level.

DETAILED DESCRIPTION:
Placebos have been in use for centuries in medical practice. However, there is continued controversy regarding their effectiveness and mechanisms of action.

The results of the study are expected to further our understanding of a widely used medical intervention, i.e., placebo, and of how to maximize its potential beneficial effect. It will also help assess the appropriateness of measuring the placebo effect by elimination, which has important ethical implications in relation to the design of randomized clinical trials.

Comparison: caffeine vs placebo. Dependent variables:4 hours area under the curve (AUC) of pharmacodynamics endpoints as well as pharmacokinetics endpoints in a subgroup.

ELIGIBILITY:
Inclusion Criteria:

* Males and nonpregnant females 18 and 40 years of age with at least high school education.

Exclusion criteria:

* Include evidence of clinically relevant deviation from normal health (such that it may affect the endpoints, make the ingestion of caffeine dangerous, or affect the pharmacokinetics/pharmacodynamics of caffeine),
* Pregnancy,
* Poor venous access,
* Hypertension (more than 140/90),
* Heart disease,
* History of panic attacks,
* Average daily caffeine consumption of more than 300 or less than 100 mg,
* Smoking,
* Alcohol abuse,
* Taking any medication other than birth control bills (including over-the-counter drugs) within one week from starting the study,
* Hypersensitivity to caffeine or related compounds,
* Hemoglobin of less than 13 gm/L, and recent (one week) acute illness

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
4 hours area under the curve (AUC) of peripheral systolic blood pressure | 4 hours
4 hours area under the curve (AUC) of energy level measured by Visual Analogue Scales. | 4 hours
4 hours area under the curve (AUC) of alertness level measured by Visual Analogue Scales. | 4 hours
4 hours area under the curve (AUC) of nausea measured by Visual Analogue Scales. | 4 hours

SECONDARY OUTCOMES:
Cmax of serum caffeine (in a subgroup) | 4 hours
Tmax of serum caffeine (in a subgroup) | 4 hours
t1/2 of serum caffeine (in a subgroup) | 14 hours
AUC of serum caffeine (in a subgroup) | 14 hours

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad M Hammami, MD, PhD, Principal Investigator — KFSH & RC, Riyadh
Locations (1):
- Center for Clinical Studies & Empirical Ethics, KFSH & RC, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Hammami MM, Al-Gaai EA, Alvi S, Hammami MB. Interaction between drug and placebo effects: a cross-over balanced placebo design trial. Trials. 2010 Nov 19;11:110. doi: 10.1186/1745-6215-11-110. PMID 21092089